CLINICAL TRIAL: NCT04762004
Title: Maternal Speech Decreases Pain Scores and Increases Oxytocin Levels in Preterm Infants During Painful Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Manuela Filippa, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 90.513
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Preterm Birth; Pain, Procedural
Keywords: Oxytocin; Maternal voice; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth; Pain, Procedural | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Crossover clinical trial with a repeated measures design. Each patient is assigned to a sequence of three treatments (maternal speech, maternal singing, and standard treatment).
Who Masked: Outcomes Assessor
Masking Description: The pain score was assessed by two blinded independent and trained coders on muted video tracks. Oxytocin analysis were performed by an external Lab, blinded to the conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maternal speech (Experimental): During the intervention, mothers were asked to speak to their preterm infants in the incubators for 5 min preceding the heel prick procedure and for the subsequent 5 min.
  Interventions: Behavioral: Maternal speech
- Maternal singing (Experimental): During the intervention, mothers were asked to sing to their preterm infants in the incubators for 5 min preceding the heel prick procedure and for the subsequent 5 min.
  Interventions: Behavioral: Maternal singing
- Standard care (Active Comparator): During the control condition (without the mother), the newborn was placed by the nurse in the incubator in the standard care conditions recommended for painful procedures (supine position, wrapped and contained by the nest).
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Maternal speech — In both intervention conditions, speaking and singing, the mothers were asked not to touch the baby but to pay close attention to his/her reactions and to modulate the voice accordingly. A nurse was present during all procedures.
  Arms: Maternal speech
Behavioral: Maternal singing — In both intervention conditions, speaking and singing, the mothers were asked not to touch the baby but to pay close attention to his/her reactions and to modulate the voice accordingly. A nurse was present during all procedures.
  Arms: Maternal singing
Behavioral: Standard care — the newborn was placed by the nurse in the incubator in the standard care conditions recommended for painful procedures (supine position, wrapped and contained by the nest).
  Arms: Standard care

SUMMARY:
Preterm infants undergo early separation from parents and are exposed to frequent painful clinical procedures, with resultant short- and long-term effects on their neurodevelopment. We aimed to establish whether the mother's voice could provide an effective and safe analgesia for preterm infants and whether endogenous oxytocin (OXT) could be linked to pain modulation. Twenty preterm infants were exposed to three conditions-mother's live voice (speaking or singing) and standard care-in random order during a painful procedure. OXT levels (pg/mL) in saliva and plasma cortisol levels were quantified, and the Premature Infant Pain Profile (PIPP) was blindly coded by trained psychologists.

DETAILED DESCRIPTION:
Preterm birth rates are continuously increasing in almost all countries, with 15 million premature infants being born every year worldwide1. Despite rapid advances in technology, the number of preterm-born children who show short- and long-term sequelae of prematurity, even before reaching school age, remains high. Around 40% of low birth weight preterm infants experience a complex spectrum of unfavourable neurodevelopmental outcomes when compared with their pairs at term. Thus, prematurity is of great concern for health policies in both low- and high-income countries. The impaired development of preterm infants is not only associated with medical factors, but it is also at least partly a consequence of the atypical early-life environment of these infants, including exposure to pain and separation from the primary caregivers.

The aim of the present work was first, to assess whether early closeness with parents during essential but painful clinical procedures could have a positive role in pain modulation in preterm infants, thus contributing to the universal right to pain relief. Second, we aimed to investigate the possible role of the oxytocinergic system in this putative pain modulation through maternal vocal contact.

In the present protocol, we introduce the effects of separation and early pain exposure as two environmental factors that are even more deleterious when concomitant, inducing short- and long-term problems in the preterm infant's development. We then suggest that there are protective effects of early closeness between parents and preterm infants in early care and, more specifically, of early vocal contact between parents and preterm infants during hospitalisation. Lastly, we discuss the role of oxytocin (OXT) as a crucial biomarker for attachment processes and in relation to brain inflammation due to stressful procedures for preterm infants in the neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

* age >29 weeks gestational age at birth,
* weight >1000 g
* stable medical condition (absence of mechanical ventilation, no additional oxygen)

Exclusion Criteria:

For infants

* no specific pathological conditions
* no genetic abnormalities

For mothers

* history of substance abuse
* mental health problems

Ages: 29 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
pain score | Immediately after the procedure
  The PIPP-R score is a cluster of physiological and behavioural measures. Physiological assessment was calculated on the heart rate and oxygen saturation levels as collected from the patient monitor by the researcher. Inter-rater reliability was assessed by three independent coders: expert coders 1 and 2 performed blinded ratings from offline muted videos and digitally recorded physiological parameters, whereas coder 3 was a trained nurse and performed a direct online rating of the scores. Higher levels of pain scores indicate higher levels of pain
oxytocin levels | Pre procedure
  Early relational experiences can persistently affect social behaviours by modifying the oxytocin system and endogenous oxytocin regulation is a potential protective mechanism for early pain perception. Higher levels of oxytocin can indicate better pain protection.
oxytocin levels | Immediately after the procedure
  Early relational experiences can persistently affect social behaviours by modifying the oxytocin system and endogenous oxytocin regulation is a potential protective mechanism for early pain perception. Higher levels of oxytocin can indicate better pain protection.

CONTACTS AND LOCATIONS:
Overall Officials: Didier M Grandjean, Professor, Study Director — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No